CLINICAL TRIAL: NCT05590390
Title: Prevalence and Impact on Quality of Life of Osteoporosis and Fragility Fractures Among SLE Patients. (FRAIL Trial)
Brief Title: Osteoporosis and Fragility Fractures Among SLE Patients. (FRAIL Trial)
Acronym: FRAIL
Status: Active, not recruiting | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Other Study IDs: 3875CESC
Record Dates: First submitted 2022-10-07; First posted 2022-10-21 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: DXA — bone densitometry at lumbar and femoral site+ morphometry (DXA),
Diagnostic Test: serum sample — serum samples for bone biomarkers ( eg. P1NP, CTX, Dkk-1, etc)
Diagnostic Test: PROs — questionnaires to investigate patients reported outcome on quality of life

SUMMARY:
The trial is designed to evaluate prevalence of fragility fracture, their impact on quality of life of SLE patients and disease or treatment variables such as steroids dosage or use of specific drugs like hydroxychloroquine, DMARDs or belimumab. Patients will perform DXA evaluation, blood tests and PROs questionnaires. Moreover, the investigators want to correlate those variables to bone turnover markers and bone metabolism modulators. A secondary aim is also to assess the fracture risk of those patients as described by FRAX and DEFRA tools.

ELIGIBILITY:
Inclusion Criteria:

* SLE fulfilling 2019 ACR/EULAR or 2012 SLICC criteria
* willing to perform DXA/ x-Ray investigation (common clinical practice)
* willing to donate blood sample
* willing to complete questionnaires
* the patients should be in a stable disease activity.

Exclusion Criteria:

* Uncontrolled endocrinological disease.
* metabolic bone disease other than osteoporosis ( e.g. Paget disease).
* celiac disease, inflammatory bowel disease or pancreatic exocrine deficiency resulting in malabsorption
* patients lacking medication history information (SLE and bone related medications).
* Have any other clinically significant abnormal laboratory value in the opinion of the investigator
* Have any intercurrent significant medical illness that the investigator considers would make the candidate unsuitable for the study.
* The patients shouldn't be enrolled during a moderate to severe flare of disease requiring an escalation of therapy ( especially glucocorticoid) - no new BILAG A or B in the last 3 months.
* Pregnant patients or during the first year after child birth.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SLE patients 18-75 years
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-12-31 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of osteoporosis | 1 visit - 1 hour
  percentage of patient with osteoporosis defined by WHO definition with T score
Prevalence of fragility fractures | 1 visit 1 hour
  percentage of patients with fragility fractures
EQ5D | 1 visit - 1 hour
  scores at questionnaire on quality of life EQ5D = EuroQol 5 dimension 5 L; (min 1-1-1-1-1, max 5-5-5-5-5 higher score worse + EQ VAS min 0, max 100 higher score better quality of life)
FACIT-F | 1 visit - 1 hour
  scores in fatigue as for questionnaire FACIT-F (Functional Assessment of Chronic Illness Therapy - Fatigue; min 0 - max 52, higher score less fatigue)
SF-36 v2 | 1 visit - 1 hour
  scores on quality of life with SF36 v2 (Short Form 36 version 2 Health Survey; min 0 - max 100, higher score better health)
HADS | 1 visit - 1 hour
  scores on mood disorder scale HADS (Health Anxiety and Depression Scale; min 0 - Max 42, higher score worse anxiety)
CQR5 | 1 visit - 1 hour
  compliance questionnaire in rheumatology 5 items; adherent - not adherent to medication)
PGA | 1 visit - 1 hour
  Patient global assessment ( VAS scale 0-10) higher score worse health
influence of SLE medication - glucocorticoid | 1 visit - 1 hour
  The population will be analyzed grouping by presence or absence of fragility fracture in relation to medications variables such as difference in cumulative corticosteroid dose (mg)
influence of SLE medication - hydroxychloroquine | 1 visit - 1 hour
  The population will be analyzed grouping by presence or absence of fragility fracture in relation to medications variables such as difference in percentage of hydroxychloroquine users.
influence of SLE medication - immunosuppressant | 1 visit - 1 hour
  The population will be analyzed grouping by presence or absence of fragility fracture in relation to medications variables such as difference in percentage percentage of immunosuppressant users
influence of SLE medication - biologics | 1 visit - 1 hour
  The population will be analyzed grouping by presence or absence of fragility fracture in relation to medications variables such as difference in percentage of percentage of biologics ( e.g. belimumab) users.

SECONDARY OUTCOMES:
Descriptive statistics of study population - 1 | 1 visit - 1 hour
  The population will be analyzed as whole and also grouping by presence or absence of fragility fracture in relation to clinical variables - SLE disease duration
Descriptive statistics of study population - 2 | 1 visit - 1 hour
  The population will be analyzed as whole and also grouping by presence or absence of fragility fracture in relation to clinical variables - SDI ( SLICC Damage index - from 0, higher score higher disease damage accrual)
Descriptive statistics of study population - 3 | 1 visit - 1 hour
  The population will be analyzed as whole and also grouping by presence or absence of fragility fracture in relation to demographic variable - Age ( years)
Descriptive statistics of study population - 4 | 1 visit - 1 hour
  The population will be analyzed as whole and also grouping by presence or absence of fragility fracture in relation to demographic variable - gender ( % females)
serum bone biomarkers - BAP | 1 visit - 1 hour
  bone alkaline phosphatase (BAP) (ug/L) level in study population and difference by fracture status
serum bone biomarkers - P1NP | 1 visit - 1 hour
  N-terminal propeptide of type I procollagen - P1NP (ng/ml) level in study population and difference by fracture status
serum bone biomarkers - CTX | 1 visit - 1 hour
  C-terminal telopeptide of type I collagen (CTX) (ng/ml), level in study population and difference by fracture status
serum bone biomarkers - PTH | 1 visit - 1 hour
  parathormone (PTH) pg/ml level in study population and difference by fracture status
serum bone biomarkers - vitamin D(OH) | 1 visit - 1 hour
  25OH vitamin D (ng/ml), level in study population and difference by fracture status
serum bone biomarkers - Sclerostin | 1 visit - 1 hour
  sclerostin (pmol/L) level in study population and difference by fracture status
serum bone biomarkers - Dkk1 | 1 visit - 1 hour
  Dkk1 (pmol/L) level in study population and difference by fracture status
serum bone biomarkers - RANKL | 1 visit - 1 hour
  RANKL (pg/ml) level in study population and difference by fracture status
serum bone biomarkers - OPG | 1 visit - 1 hour
  OPG (pg/ml level) in study population and difference by fracture status
Fracture risk calculation by FRAX tool | 1 visit - 1 hour
  FRAX fracture risk assessment ( % risk major fracture in 10 yrs)
Fracture risk calculation by DEFRA tool | 1 visit - 1 hour
  DEFRA fracture risk assessment ( % risk major fracture in 10 yrs)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Rossini, MD, PhD, Principal Investigator — AOUI Verona - University of Verona
Locations (1):
- AOUI Verona - UOC Reumatologia, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rotta D, Adami G, Galvagni I, Pistillo F, Fassio A, Gatti D, Zen M, Ravagnani V, Maiolini F, Croce J, Volpe A, Dartizio C, Benini C, Ruzzon F, Viapiana O, Rossini M, Orsolini G. Prevalence and determinants of vertebral fractures in a SLE cohort. Lupus Sci Med. 2025 Sep 14;12(2):e001508. doi: 10.1136/lupus-2025-001508. PMID 40953912